CLINICAL TRIAL: NCT01541462
Title: Weaning From Prolonged Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RML Specialty Hospital (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Amal Jubran, Attending Physician, RML Specialty Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AXJ001; 5R01NR008782 (NIH)
Record Dates: First submitted 2012-02-16; First posted 2012-03-01 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Acute Mechanical Ventilatory Failure
Keywords: mechanical ventilation; weaning; pressure support; spontaneous breathing; Long-term acute care facility; mortality
MeSH Terms: interventions — Weaning

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pressure support (Active Comparator): Patients randomized to the pressure support arm will wean using pressure support ventilation. The level of pressure support will be decreased by 2 cm H2O every 6 hours. The maximum decrement in pressure support permitted in one day will be 6 cm H2O.
  Interventions: Other: Weaning
- Spontaneous Breathing (Active Comparator): Patients randomized to spontaneous breathing arm will be disconnected from the ventilator and allowed to breathe spontaneously through the tracheostomy. Duration of the trial will be increased sequentially as tolerated.
  Interventions: Other: Weaning

INTERVENTIONS:
Other: Weaning — Decrease assistance provided by the ventilator
  Other Names: Pressure support; Spontaneous breathing

SUMMARY:
Patients requiring the use of artificial ventilation (also called mechanical ventilation) for more than 21 days account for more than 37% of all ICU costs. As such, these patients are now transferred to centers that specialize in weaning patients from the respirator; these units are referred to as long-term acute care (LTAC) facilities. Despite the increase of LTAC facilities, research on the fastest method for disconnecting the patient from the respirator is lacking. In addition, little information is available regarding the long-term survival and quality of life after a prolonged course of artificial ventilation. The purpose of this study is to determine the fastest method for disconnecting the patient from the respirator at a LTAC facility and its effect on long-term survival and quality of life.

DETAILED DESCRIPTION:
Patients requiring prolonged mechanical ventilation (defined as more than 21 days) account for more than 37% of all ICU costs. As such, these patients are now transferred to centers that specialize in weaning from mechanical ventilation, so called long-term acute care (LTAC) facilities. Despite the proliferation of LTAC facilities, research on methods for expediting weaning is lacking. In addition, little information is available regarding long-term survival and patient's perception of quality of life after a prolonged course of mechanical ventilation.

In patients receiving mechanical ventilation in an ICU, randomized trials have revealed that ventilator duration was significantly influenced by weaning methods. The two most common weaning methods are pressure support and spontaneous breathing trials. Unlike the ICU, the relative efficacy of these two techniques in weaning patients requiring prolonged ventilation at a LTAC facility is largely unknown. The aim of this proposal is to determine whether the length of time required for weaning from prolonged ventilation differs with pressure support versus spontaneous breathing trials. The second aim is to determine the long-term impact of prolonged ventilation on survival, functional status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical Ventilation for at least 21 days

Exclusion Criteria:

* Hypoxemia (oxygen saturation < 90% with fractional inspired O2 concentration > 0.40, and positive end-expiratory pressure > 5 cm H2O
* Hemodynamic instability (requiring intravenous vasoactive agents, such as dopamine > 5 mg/kg/min)
* Profound neurological deficits (large stroke)
* Documented bilateral phrenic nerve injury
* Previous admission to RML Hospital
* Life expectancy less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2000-10; Primary Completion 2010-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Weaning duration | From the first day of randomization to the day the patient was successfully weaned up to 5 days

SECONDARY OUTCOMES:
mortality | 6 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Amal Jubran, MD, Principal Investigator — RML Specialty Hospital
Locations (1):
- RML Specialty Hospital, Hinsdale, Illinois, United States

REFERENCES:
- [Derived] Jubran A, Grant BJ, Duffner LA, Collins EG, Lanuza DM, Hoffman LA, Tobin MJ. Effect of pressure support vs unassisted breathing through a tracheostomy collar on weaning duration in patients requiring prolonged mechanical ventilation: a randomized trial. JAMA. 2013 Feb 20;309(7):671-7. doi: 10.1001/jama.2013.159. PMID 23340588